CLINICAL TRIAL: NCT03449303
Title: Essential Oils Effect on Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer: A Mixed Methods Study
Brief Title: Chemotherapy-Induced Peripheral Neuropathy-Essential Oil Intervention
Acronym: CIPN-EOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: American Holistic Nurses Association (Unknown); American Nurses Foundation (Other); Ananda Apothecary (Unknown); The Jojoba Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1028595
Record Dates: First submitted 2018-01-08; First posted 2018-02-28 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Peripheral Neuropathies
Keywords: breast cancer; CIPN; Pain; QOL; Essential Oils
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Intervention Model Description: The study design uses a randomized, single-blind, placebo-controlled quantitative (QUAN) strand paralleled by a photovoice methodology qualitative (QUAL) strand.
Who Masked: Participant
Masking Description: Participants will be seen in two separate clinic rooms. Intervention and placebo will have identical packaging and labeling with the addition of an A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI (Active Comparator): 10% dilution of Curcuma longa, Piper nigrum, Pelargonium asperum, Zingiber officinale, Mentha x piperita, and Rosmarinus officinalis ct. cineole in Simmondsia chinensis
  Interventions: Other: EOI
- Placebo (Placebo Comparator): Simmondsia chinensis
  Interventions: Other: Placebo

INTERVENTIONS:
Other: EOI — Topically-applied oil
  Arms: EOI
Other: Placebo — Topically-applied oil
  Arms: Placebo

SUMMARY:
This study will evaluate an oil blend with active ingredients for the reduction in chemotherapy-induced peripheral neuropathy in people with breast cancer. Half of the participants will receive the oil blend with active ingredients and the other half will receive a placebo (an oil blend with no active ingredients). One-fourth of the people will also take pictures of their life with chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a painful, debilitating consequence of cancer treatment and is considered the most adverse of non-hematologic events. Current pharmacological approaches to reduce CIPN symptoms can be ineffective and cause adverse effects.

Constituents of this oil blend moderate pain signal transmission through non-competing inhibition of 5-HT, AchE, and Substance P, along with antagonism of TRPA1 and TRPV1. This study will test the hypothesis that an oil blend reduces CIPN symptoms and improves quality-of-life (QOL) in breast cancer patients. The Human Response to Illness model is used to underpin a convergent-nested-parallel mixed-methods design with intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer
* chronic CIPN symptoms in one or both lower extremities
* three months or greater since last chemotherapy treatment
* mean SF-MPQ-2 score of greater than or equal to three
* a prognosis of greater than six months

Exclusion Criteria:

* non-English-speaking
* blindness
* pregnancy
* breastfeeding
* allergy to EOI or Peru balsam (cross-allergen)
* illegal substance usage
* history of severe skin reactions
* non-intact skin on lower extremities
* history of lower extremity trauma or amputation
* current use of aromatherapy/Essential Oils
* asthma or reactive airway disease triggered by constituents of EOI
* history of mental illness or chronic depression
* the following co-morbidities: G6PD deficiency, inherited peripheral neuropathy, active herpes varicella-zoster, herpes simplex virus, alcoholic neuropathy, repetitive stress or entrapment neuropathy, peripheral vascular disease, and multifocal mononeuropathy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | baseline and weekly for 6 weeks
  A 22-item self-report pain intensity (over past week) peripheral neuropathy questionnaire. Each item is scored from 0 -10 (0 is no pain and 10 is the worst possible pain), a mean score is obtained, yielding a mean score between 0 and 10.

SECONDARY OUTCOMES:
Visual Analogue Scale - Pain (VAS) | Baseline and daily for 6 weeks
  A 10 cm horizontal line with a 0 (no pain) on the far left and 10 (worst possible pain) on the far right. Participants rate current pain intensity by drawing a mark on the line. Pain intensity is obtained by measuring from the 0 to the participant's mark on the line, yielding a score from 0 to 10. Daily pain scores will be averaged for a weekly mean.
Quality of Life Adult Cancer survivor (QLACS) | Baseline, week four and week seven
  The QLACS consists of 47 questions in two domains (generic and cancer-specific). The questionnaire offers respondents the following choices: 1=never, 2=seldom, 3=sometimes, 4=about as often as not, 5=frequently, 6=very often, and 7=always, yielding a total score of between 0 to 350. A mean score will be used.
Quality of Life: Chemotherapy-Induced Peripheral Neuropathy-20 (QOL:CIPN20) | Baseline, week four and week seven
  The QOL: CIPN20 consists of 20 questions represented by three scales: autonomic symptoms and functioning, sensory, and motor. Participants are to rate symptoms over the past week as 1=not at all, 2=a little, 3=quite a bit, and 4=very much. Items are scored per scale as a higher score = worse, yielding a total score of between 0 and 100. A mean score will be used.

OTHER OUTCOMES:
Sleep-related questions | Baseline, week four and week seven
  The following two questions are exploratory: In the past seven days, how many times have you slept through the night? In the past seven days, how many times did your pain wake you from sleep? If pain woke you from sleep, please describe your experience. If anything other than pain woke you from sleep, please list. Neither QOL questionnaire also address sleep. The answers to these questions will be integrated into QOL data.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Zadinsky, PhD, Study Chair — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No